CLINICAL TRIAL: NCT02248558
Title: Crowdsourcing Versus Conventional HIV Testing Promotion: A Noninferiority Randomized Controlled Trial to Evaluate Promoting First-Time HIV Testing Among MSM and Transgender Individuals in China
Brief Title: Spurring Innovation to Promote HIV Testing: An RCT Evaluating Crowdsourcing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Social Entrepreneurship to Spur Health (Other); University of California, San Francisco (Other); London School of Hygiene and Tropical Medicine (Other); Guangdong Provincial Centers for Skin Diseases and STI Control (Unknown)
Responsible Party: Principal Investigator, Joseph Tucker, MD, PhD, MA, Assistant Professor of Medicine, Director of UNC Project-China, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: 14-1865
Record Dates: First submitted 2014-09-17; First posted 2014-09-25 (Estimated); Results first posted 2016-12-20 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: HIV
Keywords: Contest; Crowdsourcing; Innovation; Randomized controlled trial; China; Social entrepreneurship

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional video (Active Comparator): This arm will receive a one-minute conventional video promoting HIV test uptake.
  Interventions: Behavioral: Conventional Video
- Crowdsourced video (Experimental): This arm will receive a one-minute crowdsourced video promoting HIV test uptake.
  Interventions: Behavioral: Crowdsourced Video

INTERVENTIONS:
Behavioral: Conventional Video — Participants will watch a one minute video whose purpose is to increase HIV testing uptake. This video was created by a local CDC via direct CDC funding and internal guidance and development.
  Arms: Conventional video
Behavioral: Crowdsourced Video — Participants will watch a one minute video whose purpose is to increase HIV testing uptake. This video was the winner in a crowdsourced video contest hosted in China. CBOs all submitted their own independently designed and funded videos.
  Arms: Crowdsourced video

SUMMARY:
Crowdsourcing may be a powerful tool to spur the development of innovative videos to promote HIV testing among key populations such as men who have sex with men (MSM) and transgender (TG) individuals. The purpose of this randomized controlled trial is to compare the effect of a crowdsourced video and a conventional video on first-time HIV testing among MSM and TG in China. The crowdsourced video was developed using an open contest, formal transparent judging, and an incentive of marketing promotion. The hypothesis is that a crowdsourced video will be equivalent (within a margin of 3%) to a conventional video in terms of self-reported first-time HIV testing within 3-4 weeks of watching the video.

ELIGIBILITY:
Inclusion Criteria:

* Born biologically male or identify as transgender
* 16 years or older
* Lifetime anal sex with another man
* Providing informed consent and active mobile phone number

Exclusion Criteria:

* HIV-infected
* HIV-tested ever in the past

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 721 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Tucker, Principal Investigator — UNC Project-China
Locations (1):
- UNC Project-China, Guangzhou, China

REFERENCES:
- [Derived] Wang C, Mollan KR, Hudgens MG, Tucker JD, Zheng H, Tang W, Ling L. Generalisability of an online randomised controlled trial: an empirical analysis. J Epidemiol Community Health. 2018 Feb;72(2):173-178. doi: 10.1136/jech-2017-209976. Epub 2017 Nov 28. PMID 29183956
- [Derived] Tang W, Han L, Best J, Zhang Y, Mollan K, Kim J, Liu F, Hudgens M, Bayus B, Terris-Prestholt F, Galler S, Yang L, Peeling R, Volberding P, Ma B, Xu H, Yang B, Huang S, Fenton K, Wei C, Tucker JD. Crowdsourcing HIV Test Promotion Videos: A Noninferiority Randomized Controlled Trial in China. Clin Infect Dis. 2016 Jun 1;62(11):1436-1442. doi: 10.1093/cid/ciw171. Epub 2016 Apr 29. PMID 27129465
- See also: Social Entrepreneurship for Sexual Health — http://www.seshglobal.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conventional Video | Crowdsourced Video
Started | 369 | 352
Completed | 317 | 307
Not Completed | 52 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Video | Crowdsourced Video | Total
Number analyzed (Participants) | 369 | 352 | 721
Age, Customized [Count of Participants; unit: Participants]
  16-20 | 114 | 120 | 234
  21-25 | 130 | 136 | 266
  26-30 | 62 | 50 | 112
  31-35 | 38 | 28 | 66
  >35 | 27 | 18 | 45
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 351 | 334 | 685
  Transgender | 18 | 18 | 36
Education [Count of Participants; unit: Participants]
  High School or below | 105 | 108 | 213
  College | 239 | 231 | 470
  Graduate Education | 25 | 13 | 38
Annual Income (SD) [Count of Participants; unit: Participants]
  <3000 | 128 | 113 | 241
  3000-6000 | 102 | 104 | 206
  6001-9500 | 85 | 84 | 169
  9501-15000 | 38 | 37 | 75
  >15000 | 16 | 14 | 30
Marital status [Count of Participants; unit: Participants]
  Never married | 304 | 311 | 615
  Married/Engaged | 50 | 39 | 89
  Separated/divorced/Widowed | 15 | 10 | 25
Sexual orientation disclosure [Count of Participants; unit: Participants]
  Yes | 210 | 199 | 409
  No | 159 | 153 | 312
Ever used gay mobile application [Count of Participants; unit: Participants]
  Yes | 267 | 275 | 542
  No | 97 | 71 | 168
Recent Condomless anal sex [Count of Participants; unit: Participants]
  No recent sex | 58 | 47 | 105
  Condomless anal sex | 23 | 28 | 51
  Anal sex with a condom | 57 | 58 | 115

OUTCOME MEASURES:

1. Primary Outcome: First-Time HIV Testing
Description: All individuals enrolled in the study will receive a cell phone text message three weeks later asking if they have received an HIV test. Among those individuals who do not respond to the text message, another text will be sent at four weeks after the video. We anticipate the median duration of follow-up to be approximately 3.5 weeks following the video intervention.
Time Frame: Up to 4 weeks following the video intervention
Measure: Count of Participants; unit: Participants
Groups:
- Conventional Video: This arm will receive a one-minute conventional video promoting HIV test uptake.
  Conventional Video: Participants will watch a one minute video whose purpose is to increase HIV testing uptake. This video was created by a local CDC via direct CDC funding and internal guidance and development.
  111 of 317 (35%) in the health marketing arm reported testing for HIV
- Crowdsourced Video: This arm will receive a one-minute crowdsourced video promoting HIV test uptake.
  Crowdsourced Video: Participants will watch a one minute video whose purpose is to increase HIV testing uptake. This video was the winner in a crowdsourced video contest hosted in China. CBOs all submitted their own independently designed and funded videos.
  In the crowdsourced intervention arm, 114 of 307 (37%) reported testing for HIV.
Arm/Group | Conventional Video | Crowdsourced Video
Number analyzed (Participants) | 317 | 307
Participants | 111 | 114

2. Secondary Outcome: Likelihood of HIV Testing
Description: All individuals will be asked how likely they are to test for HIV soon immediately before and after watching the videos (during enrollment). Likelihood of HIV testing will be measured on a 4-point numerical Likert scale rating scale. 0 will be "very unlikely", 1 will be "unlikely", 2 will be likely, and 3 will be very likely. The percentage of individuals who report increased likelihood of HIV testing will be reported.
Time Frame: Up to one day
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Video | Crowdsourced Video
Number analyzed (Participants) | 369 | 352
Participants
  Yes | 184 | 212
  No | 185 | 140

3. Secondary Outcome: Cost-effectiveness of Developing HIV Testing Promotional Videos
Description: Cost-effectiveness of developing the crowdsourced video compared to the conventional video
Time Frame: Up to one year
Measure: Number; unit: USD
Arm/Group | Conventional Video | Crowdsourced Video
Number analyzed (Participants) | 369 | 352
USD
  The incremental unit cost for promoting HIV testin | 238 | 131
  The incremental unit costs per newly diagnosed HIV | 799 | 415

ADVERSE EVENTS:
Arm/Group | Conventional Video | Crowdsourced Video
Serious Adverse Events (participants affected / at risk) | 0/369 | 0/352
Other Adverse Events (participants affected / at risk) | 0/369 | 0/352

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No